CLINICAL TRIAL: NCT04585568
Title: Validation and Comparison of Ballistocardiographic Biosensors and Other Hemodynamic Measures for Healthy Subjects During Different Situations
Brief Title: Validation of Ballistocardiographic Biosensors and Other Hemodynamic Measures for Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Telemedicine (Unknown); Kopera Norway (Unknown); Edwards Lifesciences (Industry); Stryker Medical (Industry); University of the Basque Country (UPV/EHU) (Other); University of Stavanger (Other)
Responsible Party: Principal Investigator, Lars Wik, Principle Investigator, Oslo University Hospital
Other Study IDs: 153368
Record Dates: First submitted 2020-10-01; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Hemodynamics; Biosensors; Cardiac
Keywords: blood flow; correlations; ballistocardiography; invasive blood pressure; cardiac output; doppler eccocardiography
MeSH Terms: interventions — Biosensing Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biosensors — Measures of blood flow and preassures
  Other Names: FloTrac; Doppler eccocardiography

SUMMARY:
Ballistocardiographic (BCG) biosensors reflecting the patients' current state is established. There are few studies documenting BCG biosensors efficacy, effectiveness, and efficiency. In addition, technologies using invasive blood pressure curves and Near Infrared Regional Spectrometry (NIRS) to measure hemodynamics have been used. Using these technologies to guide clinical decisions may be an major advance for patients with acute and chronic diseases. The investigators will explore how these technologies compares to well established technologies measuring vital signs of healthy subjects. The investigators will use live continuous and non-continuous biosensor data to monitor the development of vital parameters during different scenarios. The study will document how CPD measured by biosensors, cerebral oximetry measured by NIRS, and invasive blood pressure curves measured by FloTrac™ are compared to established technologies of vital organ functionality.

Data will be measured continuously and documented simultanuously with technologies such as Doppler Echocardiography, transthoracic impedance (TTI), Electrocardiogram (ECG), invasive blood pressure [cardiac output/index (CO/CI), stroke volume/stroke volume index (SV/SVI), stroke volume variation/pulse pressure variation (SVV/PPV), systemic vascular resistance/ systemic vascular resistance index (SVR/SVRI), mean arterial pressure (MAP)], pulse oximetry (SpO2) and cerebral oximetry (rSO2). Of special interest is to document how relative heart stroke volume reflects blood flow documented by the parallel technology measures. All these measures are the key part in the study to document user friendliness, accuracy, sensitivity, specificity and correlations.

The main research question is whether adding BCG biosensor measures, cerebral oximetry and invasive blood pressure to monitor vital signs will add meaningful information to the care of patients in a situation where we are able to control all the factors that may impact these measures. The aim of the study is to document (correlation, sensitivity and specificity) how BCG biosensors perform compared to each other and to well established technologies used for monitoring blood flow, blood pressure, heart rate and respiration rate in steady state and during ambulance transport. In addition, the investigators will in a controlled manner measure how established maneuvers like Trendelenburg, hypo-/hyperventilation, and bolus of fluid influences our measures.

DETAILED DESCRIPTION:
Ballistocardiographic (BCG) biosensors collecting continuous physiological data (CPD) in real time to generate information reflecting the patients' current state is established and have become more useful in monitoring vital signs of subjects and patients. There are few studies documenting BCG biosensors efficacy, effectiveness, and efficiency. Using CPD to guide clinical decisions may be a major advance for patients with acute and chronic diseases. In addition, technologies using invasive blood pressure curves and Near Infrared Regional Spectrometry (NIRS) to measure hemodynamics have been used. This may drive the evolution from episodic to continuous patient care for these patients experiencing a severe medical event compromising blood flow. The investigators will explore how these technologies compares to well established technologies measuring vital signs of healthy subjects. In the present study the investigators will use live continuous and non-continuous biosensor data to monitor the development of vital parameters during different scenarios. The study will document how CPD measured by biosensors, cerebral oximetry measured by NIRS, and invasive blood pressure curves measured by FloTracTM are compared to established technologies of vital organ functionality.

In the present study data will be measured continuously and in phases of the study simultaneously with other well established technologies such as Doppler Echocardiography, transthoracic impedance (TTI), Electrocardiogram (ECG), invasive blood pressure [cardiac output/index (CO/CI), stroke volume/stroke volume index (SV/SVI), stroke volume variation/pulse pressure variation (SVV/PPV), systemic vascular resistance/ systemic vascular resistance index (SVR/SVRI), mean arterial pressure (MAP)], pulse oximetry (SpO2) and cerebral oximetry (rSO2). Based on this the investigators believe they will be able to pick up how dynamic differences develop. Of special interest is to document how relative heart stroke volume reflects blood flow documented by the parallel technology measures. HRV will also be evaluated in the light of other measures such as pulse, respiration, and relative stroke volume. All these measures are the key part in the study to document user friendliness, accuracy, sensitivity, specificity and correlations.

The main research question is whether adding BCG biosensor measures, cerebral oximetry and invasive blood pressure to monitor vital signs will add meaningful information to the care of patients in a situation where we are able to control all the factors that may impact these measures. The aim of the study is to document (correlation, sensitivity and specificity) how BCG biosensors perform compared to each other and to well established technologies used for monitoring blood flow, blood pressure, heart rate and respiration rate in steady state and during ambulance transport. In addition, the investigators will in a controlled manner measure how established maneuvers like Trendelenburg, hypo-/hyperventilation, and bolus of fluid influences our measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who have signed informed consent

Exclusion Criteria:

* Sick subjects at test day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Paramedic students recruited free of will.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between different measures of hemodynamics | September to December
  Calculated based on a number of hemodynamic measures listed in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Please Select, Norway

IPD SHARING:
Plan to Share IPD: Yes
Based on informed consent this will be done with those parties listed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From September 2020 to September 2025
Access Criteria: A secure sharing plattform will be used.